CLINICAL TRIAL: NCT07051200
Title: Recovery Through Inspiration, Support, and Empowerment
Acronym: RISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Joseph Guillory, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2024-0135
Record Dates: First submitted 2025-04-30; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Suicidal Ideation; Suicide Attempt; Anxiety; Depression Disorders
Keywords: Peer Support Specialist (PSS); Recovery Community Organization (RCO); Mental Health Recovery; Transitional Age Youth (TAY); UT Southwestern Medical Center; Young Adult
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Cohort A: Intervention Group Cohort B: Standard of Care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A: Intervention group with PSS and RCOs (Experimental): One on one meetings peer support specialist (PSS) for education and support. Group meetings with PSS and other participants. Qualitative and quantitative assessments.
  Interventions: Behavioral: Peer Support Services Recovery
- Cohort B: Standard of Care (No Intervention): Scheduled telephone call visit with a member of the research team. Qualitative and quantitative assessments.

INTERVENTIONS:
Behavioral: Peer Support Services Recovery — A program of mental health recovery through one-on-one and small group meetings with a PSS and RCOs for individuals recently discharged from an acute care psychiatric facility.
  Arms: Cohort A: Intervention group with PSS and RCOs

SUMMARY:
The goal of this pilot study is to test the effectiveness of a novel intervention for young adults (ages 18-27) with mental health conditions who have been released from an acute care psychiatric facility. The intervention aims to reduce suicidality, depression, anxiety, re-hospitalization, and improve mental health recovery by using outpatient services.

The current standard of care (SOC) for these patients at discharge includes a discharge plan with a list of their medications, anticipated outpatient appointments, and information on when and where to find community resources.

The intervention being tested involves the implementation of a mental health recovery education and support program, involving one-on-one and small group meetings led by Peer Support Specialists (PSS) and Recovery Community Organizations (RCO).

Participants will be assigned to either Cohort A or B for 8 weeks.

Cohort A will be the intervention group with PSS and RCOs.

* Weeks 1-4: One-on-one meetings with PSS for education and support. Assessments will be completed at weeks 2 and 4.
* Weeks 5 and 7: One-on-one meetings with PSS for education and support.
* Week 6 and 8: Group meetings with PSS and other participants from RCOs. Assessments will be completed during these weeks.

Cohort B will be the SOC group with no PSS or RCOs.

* Weeks 1-4: Weekly check in phone calls with a member of the research team. Assessments will be completed at weeks 2 and 4.
* Weeks 5-8: Check in phone calls with a member of the research team every other week. Assessments will be completed at weeks 6 and 8.

Data collected from participant assessments, adherence to medication, and re-admittance to a psychiatric facility will be used to compare the intervention to the SOC.

DETAILED DESCRIPTION:
Purpose

* This is a pilot study to test the effectiveness of a novel intervention aimed at reducing the incidences of suicidality, depression, anxiety, re-hospitalization rates, and improving mental health recovery by utilizing outpatient services, and medication adherence for young adults (18-27) with mental health conditions verses the standard of care (SOC) at discharge which only provides a discharge plan with a list of their medication(s), anticipated outpatient appointment(s), and corresponding information on when and where to find community resources.
* The intervention will use peer support specialist (PSS) and recovery community organizations (RCO) aimed at improving knowledge, awareness, and utilization of recovery and wellness programs for those patients recently discharged from an acute psychiatric treatment facility.

Objectives

* Implement a program of mental health recovery education and support through one-on-one and small group meetings with a PSS and RCOs for individuals recently discharged from an acute care psychiatric facility to determine the effectiveness of: Reduction of suicidality, depression, anxiety, re-hospitalization rate AND Improvement in mental health recovery by participating in outpatient services, and medication adherence.
* Determine if peer-led interventions improve knowledge, awareness, and utilization of recovery and wellness programs and support.

Endpoints

* Determine the efficacy of peer-led, one-on-one and group sessions vs standard of care (SOC) based on responses to assessments, adherence to medication, and re-admittance to a psychiatric facility.
* Determine if there is a difference in outcome based on demographics (age, race, ethnic background, diagnosis, public vs private insurance, and zip code)

Study Design This is a 1:1 randomized, 8-week interventional study that will include an orientation session and a collection of baseline data. At the conclusion of the orientation session, subjects will be randomly assigned to Cohort A or B. Target recruitment is 40 subjects for this pilot study; 20 subjects in cohort A and 20 in cohort B. At the conclusion of the study, both groups will be provided a list of resources for therapy, outpatient psychiatry providers/services, RCOs, local emergency departments and inpatient psychiatric facilities.

Cohort A - Intervention group with PSS and RCOs

* Weeks 1-4: one-on-one meetings with peer support specialist (PSS) for education and support. Qualitative and quantitative assessments completed at weeks 2 and 4
* Weeks 5-8: Biweekly (every other week) of one-on-one meetings with PSS for education and support. Biweekly group meetings with PSS and other participants. Qualitative and quantitative assessments completed at weeks 6 and 8

Cohort B - SOC group with no PSS or RCOs; participants are responsible for finding resources or group support by following the information provided at discharge

* Weeks 1-4: Weekly check-in phone calls with a member of the research team. Qualitative and quantitative assessments completed at weeks 2 and 4 (completed during phone call check in)
* Weeks 5-8: Biweekly (every other week) check-in phone calls with a member of the research team. Qualitative and quantitative assessments completed at weeks 6 and 8 (completed during phone call check in).

ELIGIBILITY:
Inclusion Criteria:

* Chief complaint of suicidal ideation, suicide attempt, depression, and/or anxiety
* discharged from inpatient care or from emergency department
* men and women ages 18-27

Exclusion Criteria:

* primary diagnosis of: substance use disorder, schizophrenia spectrum, intellectual development disorder, autism spectrum disorder (level II or III)

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in suicidal ideation | Weeks 2, 4, 6, and 8.
  The intervention in this study will use peer support specialist (PSS) and recovery community organization (RCO) programs to improve knowledge, awareness, and utilization of recovery and wellness programs.
  Connecting patients with a PSS and recovery organizations has been associated with an improvement in patient outcomes - including a change in the incidences of suicide/attempted suicide.
  Changes in suicide ideation and consequently the mortality from suicide will be determine by administrating the Columbia Suicide Severity Rating Scale (C-SSRS) using both the baseline and since last visit assessment versions. Scoring of the assessment indicates severity.
  Changes is scores will be analyzed to determine the effectiveness of the intervention.

SECONDARY OUTCOMES:
Changes in symptoms associated with anxiety and depression | Weeks 2, 4, 6 and 8
  A reduction of anxiety and depression symptoms and rates of occurrence will be measured using the following standardized assessments:
  1. Generalized Anxiety Disorder (GAD) 7 - a widely used screening tool for assessing the severity of generalized anxiety disorder (GAD) and consists of 7 items that evaluate anxiety symptoms over the past two weeks.
  2. The Patient Health Questionnaire (PHQ) - a self reported inventory used as a screening and diagnostic tool for depression.
  Responses on each assessment at each time point specified in the protocol, will be reviewed for changes (as indicating by the scoring of frequency or severity) to determine the efficacy of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Guillory, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
At this time - there is no intention of sharing individual participant data as this is a pilot study, and due to the relatively small number of participants, any data that is shared or published will be in aggregate.

REFERENCES:
- [Background] Davidson L, Bellamy C, Guy K, Miller R. Peer support among persons with severe mental illnesses: a review of evidence and experience. World Psychiatry. 2012 Jun;11(2):123-8. doi: 10.1016/j.wpsyc.2012.05.009. PMID 22654945
- [Background] Walker G, Bryant W. Peer support in adult mental health services: a metasynthesis of qualitative findings. Psychiatr Rehabil J. 2013 Mar;36(1):28-34. doi: 10.1037/h0094744. PMID 23477647
- [Background] Lyons N, Cooper C, Lloyd-Evans B. A systematic review and meta-analysis of group peer support interventions for people experiencing mental health conditions. BMC Psychiatry. 2021 Jun 23;21(1):315. doi: 10.1186/s12888-021-03321-z. PMID 34162340
- See also: Related Info — https://www.healthyntexas.org/indexsuite/index/mentalhealth?localeType=3&parentLocale=2631
- See also: SAMSHA's working definition of recovery — https://library.samhsa.gov/sites/default/files/pep12-recdef.pdf